CLINICAL TRIAL: NCT00895427
Title: A Cross-Sectional Study Comparing Noninvasive Skin Fluorescence to Coronary Artery Calcification Measured by Rapid Computed Tomography
Brief Title: A Study Comparing Skin Fluorescence to Coronary Artery Calcification
Acronym: CACS
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Collaborators: New Mexico Heart Institute, PA (Other)
Responsible Party: Sponsor
Other Study IDs: VL-2709
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes; Coronary Artery Calcification
Keywords: Coronary artery calcification
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (12):
- 1: Male ages 45-54, without diabetes, CAC score from 0 to >1000
- 2: Male ages 55-64, without diabetes, CAC score from 0 to >1000
- 3: Male ages 65+, without diabetes, CAC score from 0 to >1000
- 4: Male ages 45-54, with diabetes and CAC score from 0 to >1000
- 5: Male ages 55-64, with diabetes, CAC score from 0 to >1000
- 6: Male ages 65+, with diabetes, CAC score from 0 to >1000
- 7: Female ages 50-59, without diabetes, CAC score from 0 to >1000
- 8: Females ages 60-69, without diabetes and CAC score from 0 to >1000
- 9: Females ages 70 +, without diabetes, CAC score from 0 to >1000
- 10: Female ages 50- 59, with diabetes, CAC score from 0 to >1000
- 11: Female ages 60-69, with diabetes, CAC score from 0 to >1000
- 12: Female age 70+, with diabetes, CAC score from 0 to >1000

SUMMARY:
This study examines the relationship between the SCOUT DM device and coronary artery calcification as determined by rapid computed tomography in patients at risk for coronary heart disease.

DETAILED DESCRIPTION:
This is a cross-sectional, single site, cohort screening trial. The correlation between the measured skin fluorescence and the CACS will be determined using a design that includes stratification by gender, subject age and subject CAC score. This design requires a single patient visit to the clinical site and a single measurement on the SCOUT device.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 45 years or females ≥ 50 years old that have had a coronary artery calcification score determined by rapid computed tomography at the clinical site within the last six months.

Exclusion Criteria:

* Receiving investigational treatments
* Psychosocial issues that interfere with an ability to follow study procedures
* Known to be pregnant
* Receiving dialysis or having known renal compromise
* Scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
* Recent or current oral steroid therapy or topical steroids applied to the left forearm
* Current chemotherapy, or chemotherapy within the past 12 months
* Receiving medications that fluoresce*
* Known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are sorted into the follwoing categories for age (years): men:45-54,55-64,65+, women: 50-59, 60-69, 70+. In addition, subjects will be sorted into the follwoing categories for CACS:0-10, 11-100, 101-400, 401-1000, >1000 and absence/presence of diagnosed diabetes (type 1 or type 2)
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Maynard, MS, Study Director — VeraLight, Inc.
Locations (1):
- New Mexico Heart Institute, Albuquerque, New Mexico, United States